CLINICAL TRIAL: NCT00385333
Title: A Novel Non-Invasive In Vivo Imaging System to Measure Retinal Metabolism
Brief Title: Metabolic Mapping to Measure Retinal Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 060252; 06-EI-0252
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-16

CONDITIONS: Macular Degeneration; Diabetic Retinopathy; Hippel-Landau Disease; Mitochondria
Keywords: Mitochondrion; Retina; Mitochondria; Metabolism; In Vivo Imaging; Age-Related Macular Degeneration; AMD; Diabetic Retinopathy; DR; Hippel-Lindau Disease; VHL
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; von Hippel-Lindau Disease

INTERVENTIONS:
Procedure: Feasibility Study - Imaging System

SUMMARY:
This study will test whether a new non-invasive technique can quickly and precisely measure retinal metabolism (the amount of energy retinal cells use). The retina is the part of the eye that sends information to the brain.

Participants in current NEI studies who have age-related macular degeneration (AMD), diabetic retinopathy, or von Hippel-Landau disease may be eligible for this study. Healthy volunteers will participate as controls. Patients with AMD must be 60 years of age or older; those with VHL disease or diabetic retinopathy must be 18 or older.

Participants undergo the tests and procedures required in the NEI study in which they previously enrolled. In addition, for the current study, they undergo metabolic mapping. For this procedure, the subject's eyes are dilated, and different amounts of low-level light are shone into the eye to see how different cells respond with changes in metabolism. Measurements are taken while the subject breathes room air and while he or she breathes medical grade oxygen for about 1 minute. The entire procedure takes about 15 minutes.

DETAILED DESCRIPTION:
Background. Alterations in retinal metabolism are associated with blinding conditions and vision loss. We propose to apply a non-invasive in vivo retinal imaging system to investigate key physiologic processes affecting retinal metabolism. The imaging system is designed to quantify and characterize the topology of retinal metabolism in 3-dimensional space across 40--130 picosecond time periods and allows dynamic measurement of physiologically relevant events.

Objectives. The primary objectives of our study are to: (1) evaluate the utility of this system in a clinical setting; and (2) examine variation in retinal metabolism within retinal cell subtypes under environmental conditions optimized to support this metabolism. The working hypothesis of our first objective is that the imaging system will be easily and efficiently implemented in a clinical setting and will yield stable and repeatable results. The working hypothesis for our second objective is that people with or at high risk for progression to sight threatening retinal disease will exhibit different metabolic profiles than an age- and sex-matched disease-free comparison group. Their peers with less severe disease may exhibit differences with severe diseased and non-diseased groups. The long-term goal of the project is to address the following research questions: Are metabolic profiles generated by the imaging system effective for determining presence and severity of retinal diseases?; and if so, are these metabolic profiles useful in identifying people at risk for progression to sight threatening forms of retinal diseases?

Study Population. We will first apply the systems in 3 groups of 10 people exhibiting a range of severity in retinal diseases that influence retinal metabolism; these diseases are: age-related macular degeneration (AMD); diabetic retinopathy (DR); and von-Hippel-Lindau (VHL) disease.

Design. Cross-sectional sampling design. If the system yields accurate, stable, and repeatable results it will be applied in longitudinal studies to evaluate prognostic utility for estimating the risk of progression to sight-threatening AMD, DR, or VHL disease.

Outcome Measures. The magnitude and 3-D topographic profile of fluorescence anisotropy values across physiologically meaningful time periods for a 20 degree field centered on the macula. Fluorescence anisotropy of our system provides a measure of retinal metabolism.

ELIGIBILITY:
* INCLUSION CRITERIA:

GENERAL INCLUSION CRITERIA:

1. Ability and willingness to provide informed consent.
2. Presence of a natural lens in the study eye(s).
3. Media clarity, pupillary dilation, and cooperation sufficient to perform measurements.
4. All participants will have the ability to read with at least 1 eye

AMD-SPECIFIC INCLUSION CRITERIA:

Participants will range from those with no AMD and little or no drusen in either eye through end stage AMD (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in one eye. Participants will be classified with the AREDS System for Classifying Age-Related Macular Degeneration and will exhibit a range of severities of AMD with at least half exhibiting unilateral advanced AMD (geographic atrophy or neovascular AMD) and half at high risk of progression. Inclusion criteria are as follows:

1. A diagnosis of AMD. We will use AREDS criteria and diagnostic scales for the definition of AMD.
2. Men and women aged 60 years or older. Children are not included because AMD (by definition) is a disease afflicting adults.
3. Eligible participants may have no evidence of AMD with little or no drusen in either eye, or may have any stage of AMD through end stage (geographic atrophic, retinal pigment epithelial detachment, or other signs of neovascular/exudative disease) in one eye.

DR-SPECIFIC INCLUSION CRITERIA:

1. People with DR will be classified with the modified ETDRS scale; participants will have a range of severities of DR, with at least half classified in the severe non-proliferative DR category (SNPDR). Efforts will be made to recruit people with unilateral SNPDR.
2. Participants will be men and women aged 18 years or older with diagnosis of diabetes mellitus (type 1 or type 2). Any one of the following will be considered sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes.
   * Current regular use of oral antihyperglycemia agents for the treatment of diabetes.
   * Documented diabetes by ADA guidelines.

VHL-SPECIFIC INCLUSION CRITERIA:

1. Participants will be men and women aged 18 years or older with a genetic confirmation of VHL-disease.
2. People with VHL disease exhibit a range of retinal lesions from none to severe.

EXCLUSION CRITERIA:

GENERAL EXCLUSION CRITERIA:

1. Cataract surgery in the study eye.
2. Glaucoma with evidence of optic nerve damage.
3. Chronic requirement for any systemic or ocular medication for other eye diseases other than AMD, DR, or VHL-disease.
4. Presence of implanted medical devices that may be affected by electromagnetic frequency (EMF) emissions. Although our equipment is CE or UL rated for EMF emissions it would be prudent to exclude people with implanted pacemakers, neural stimulators, and insulin pumps.
5. Arrhythmia as indicated in medical records, as this may result in instability in measurements.
6. History of seizures. The scanning mechanism of the system operates at 12 Hz, which may induce a seizure (n.b. a 12Hz scan rate is used in the Heidelberg HRTII and HRA).
7. Presence of chronic obstructive pulmonary disease (COPD) or other lung disease that might make breathing 100% O2 unsafe.
8. Ocular disease (other than AMD, DR, or VHL) that confounds assessment of the retina. These include but are not limited to central serous choroidopathy, optic atrophy, retinal vein occlusion, active uveitis, significant explained or unexplained visual field loss, or any other type of retinopathy or retinal degeneration.
9. Vitreous hemorrhage.
10. History of renal failure requiring dialysis or renal transplant.
11. Existing condition that in the opinion of the investigator would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09-29; Primary Completion 2008-06-01 (Actual); Study Completion 2010-09-16 (Actual)

PRIMARY OUTCOMES:
Fluorescence anisotropy

SECONDARY OUTCOMES:
The difference in fluorescence anisotropy values within subjects under room air and 100% oxygen exposure (one minute exposure time).

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Beatty S, Koh H, Phil M, Henson D, Boulton M. The role of oxidative stress in the pathogenesis of age-related macular degeneration. Surv Ophthalmol. 2000 Sep-Oct;45(2):115-34. doi: 10.1016/s0039-6257(00)00140-5. PMID 11033038
- [Background] Nyengaard JR, Ido Y, Kilo C, Williamson JR. Interactions between hyperglycemia and hypoxia: implications for diabetic retinopathy. Diabetes. 2004 Nov;53(11):2931-8. doi: 10.2337/diabetes.53.11.2931. PMID 15504974